CLINICAL TRIAL: NCT04009356
Title: Impact of Bariatric Surgery in Patients With Morbid Obesity. Prospective Study With Comparison Before and After
Brief Title: Impact of Bariatric Surgery in Patients With Morbid Obesity
Acronym: IVBIA
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Laurent BRUNAUD, Principal investigator, Professor of Surgery, Central Hospital, Nancy, France
Other Study IDs: ID-RCB:2019-A01229-48
Record Dates: First submitted 2019-06-20; First posted 2019-07-05 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Obesity, Morbid; Anal Incontinence; Image, Body
MeSH Terms: conditions — Obesity, Morbid; Encopresis | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bariatric surgical procedures — gastric bypass, sleeve, banding,biliopancreatic diversion

SUMMARY:
The main objective is to compare the prevalence of anal incontinence (AI) before and after bariatric surgery in obese patients.

Inclusion: Patients who are scheduled for a bariatric surgical procedure after a multidisciplinary evaluation for about 1 year (following french national recommendations).

Primary objective: After inclusion, all patients will fill in a specific self-questionnaire evaluating AI (PFDI-20 score) before surgery and at 6 months after surgery.

Investigators will evaluate the prevalence of anal incontinence before and at 6months after surgery using this PFDI- 20 score.

In those patients with preoperative anal incontinence (only in patients with 3 positive answers to question n°9,10, and 11 of PFDI-20 score self-questionnaire), a pelvic MRI will be performed before and at 6 months after surgery. Consequently, no further imaging exam will be performed in patients without preoperative anal incontinence (less than 3 positive answers to question n°9,10, and 11),

Secondary objectives:

* to evaluate the AI severity variation before and at 6 months after bariatric surgery regarding the percentage of postoperative weight loss.
* to compare the quality of life (PFIQ-7 score) related to AI day before and at 6 months after bariatric surgery.

DETAILED DESCRIPTION:
This study is proposed to all obese patients evaluated for potential bariatric surgery during a multidisciplinary evaluation for about 1 year following current french national recommendations.

Demographics are collected from medical records (age, sex, weight, height, diabetes, sleep apnea syndrome, hypertension, lipid disorders, distal neuropathy, depression, number of pregnancies, history of vaginal delivery, traumatic delivery, caesarean section, hysterectomy, urinary incontinence surgery, proctologic surgery, presence of rectal prolapse (operated or not), cholecystectomy, digestive resection, menopause, history of urinary or fecal or gaseous leakage, current treatments, tobacco consumption, diet.

Data are collected by self-questionnaire to all included patient during the preoperative consultation (about 6 weeks before bariatric surgery) and during the 6-months postoperative clinical visit scheduled during the regular follow-up.

ELIGIBILITY:
Inclusion Criteria:

* BMI>40 kg/m2
* BMI> 35 kg/m2 with comorbidity ( high blood pressure, diabetes, dyslipidemia, sleep apnea syndrome)

Exclusion Criteria:

* anal incontinence due to chronic diarrhea
* transit constipation
* peripheral neuropathy (diabetes ...)
* patient opposition
* any previous bariatric surgical procedure
* any pelvic surgical procedure performed during the study period (between preoperative and postoperative period at 6 months)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for a bariatric surgical procedure after a multidisciplinary evaluation for about 1 year (following HAS national recommendations).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of anal incontinence before and after bariatric surgery (%) | at 6 month postoperatively
  PFDI-20 score (pelvic floor distress inventory) from zero to 12 (0: no incontinence and 12: severe incontinence)

SECONDARY OUTCOMES:
Severity of anal incontinence before and after surgery (score) | at 6 month postoperatively
  PFDI-20 score (pelvic floor distress inventory) from zero to 12 (0: no incontinence and 12: severe incontinence)
quality of life related to anal incontinence (score) | at 6 month postoperatively
  PFIQ-7 (pelvic floor impact questionnaire) from 0 to 16 (0: no incontinence and 16: severe incontinence)
Pelvic imaging (MRI) | before and at 6 month postoperatively
  MRI

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy - Département Chirurgie Viscérale, Métabolique et Cancérologique CVMC (7ème étage), Nancy, France